CLINICAL TRIAL: NCT04282005
Title: Metabolic Surgery for the Treatment and Understanding of Non-Alcoholic Steato-Hepatitis (NASH): Weight-Dependent and Weight-Independent Effects
Brief Title: Metabolic Surgery for Steato-Hepatitis
Acronym: MeSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 267076
Record Dates: First submitted 2019-09-20; First posted 2020-02-24 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2019-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD); Non-Alcoholic Steato-Hepatitis (NASH)
Keywords: Metabolic Surgery; Bariatric Surgery; NASH; Diabetes; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Obesity | interventions — Metabolic Networks and Pathways; Bariatric Surgery; Diet

STUDY DESIGN:
Intervention Model Description: This study's population includes patients with severe obesity and non-alcoholic fatty liver disease who are eligible for bariatric surgery and are on the waiting list for either Roux en Y gastric bypass or sleeve gastrectomy at King's College Hospital.
  Main outcome measures will include several markers of inflammation and liver fibrosis assessed in plasma samples and Fine Needle Aspiration of the liver. Secondary outcome measures will include novel markers of cardiovascular risk, bile acids as well as standard markers of metabolic disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery group (Experimental): Fourteen patients who meet study criteria will be assigned to the study group and will undergo surgery; 7 RYGB and 7 SG, as planned for their standard care.
  Interventions: Procedure: Metabolic/Bariatric surgery
- lifestyle and diet (Active Comparator): Fourteen patients matched to the surgery group for age, gender, BMI, diabetes status, and NALFD score will undergo additional lifestyle interventions, dietary counselling and or meal replacement by a dietician aimed at inducing at least a 5-7% weight reduction, prior to their surgery (while on the waiting list for surgery).
  Interventions: Other: Lifestyle and Diet

INTERVENTIONS:
Procedure: Metabolic/Bariatric surgery — Patients will undergo surgery; 7 RYGB and 7 SG, as planned for their standard care.
  Arms: surgery group
Other: Lifestyle and Diet — Patients will be provided with a lifestyle interventions including dietary counselling choosing between a Low-Calorie Diet or a Meal Replacement Diet.
  Arms: lifestyle and diet

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is associated with obesity and type 2 diabetes mellitus (T2DM) and is characterised by excess liver fat on imaging or histology. NAFLD affects up to 25% of the Western population. It's more aggressive form is non-alcoholic steatohepatitis (NASH) characterised by cell injury, inflammation and fibrosis, and is associated with increased mortality from liver and cardiovascular disease. Currently, there is no specific treatment for NASH. Diet and exercise-induced weight loss remain the only recommended options. However, maintaining weight loss in the long term is difficult. There is therefore a significant unmet need for effective therapy in patients with NASH that can address the underlying mechanisms of disease. Although preliminary observational evidence suggests that bariatric/metabolic surgery, especially RYGB can improve NASH, no controlled trials to date has confirmed the efficacy of surgery compared to standard weight loss programs. Also, while animal and clinical studies have shown that bariatric surgery exerts weight-independent effects on glucose metabolism, it is yet unknown if the observed effects of bariatric/metabolic surgery on NASH are due to weight loss alone or result from additional, weight-independent mechanisms, like in the case of T2DM. If the effect of surgery on inflammation, liver fibrosis and other mechanisms of cardiometabolic risk were found to be independent on weight reduction, there would be profound and far-reaching implications for both the treatment and the understanding of NASH, cardiovascular disease and obesity-related cancers.

This project will investigate the hypothesis that, similarly to surgical control of diabetes, bariatric/metabolic surgery can also exert weight-independent effects on mechanisms of disease in NAFLD/NASH (i.e. influence on lowgrade inflammation and markers of fibrosis)

DETAILED DESCRIPTION:
This study's population includes patients with severe obesity (BMI >35kg/m2 or >32.5. kg/m2 if patient of South Asian, Caribbean or Black ethnicity) and non-alcoholic fatty liver disease (NAFLD) who are eligible for bariatric/metabolic surgery and are on the waiting list for either Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG) at King's College Hospital. Patients who meet study criteria will be assigned to the study groups as described below:

1. Surgery Group: Fourteen patients who meet study criteria will be assigned to the study group and will undergo surgery; 7 RYGB and 7 SG, as planned for their standard care.
2. Lifestyle Intervention Group: Fourteen patients matched to the surgery group for age, gender, BMI, diabetes status, and NAFLD score will undergo additional lifestyle interventions, dietary counselling (either a meal replacement diet or a low calorie diet) by a dietician aimed at inducing at least a 5-7% weight reduction, prior to their surgery (while on the waiting list for surgery).

Each participant in both the surgery and lifestyle intervention group will then attend the baseline visit.

At the baseline visit the participant will undergo a metabolic lab panel from bloods already provided to the clinic. This visit will also involve the clinical team performing an ultrasound-guided fine needle aspiration (FNA) of the liver. The fine needle aspiration will involve inserting a small needle through the skin to take a small sample of cells from the liver. It will be carried out in the Institute of Liver Studies at King's College Hospital. The clinical research team will also access the participants medical record to collect data from your medical history including weight, height, body mass index (BMI) and previous FibroScan®. Additionally, a saliva swab, urine and stool sample will be collected.

A subgroup of patients (6 participants in the Lifestyle Intervention Group, 6 undergoing RYGB, 6 undergoing SG) will undergo a mixed meal test (MMT) to investigate changes in meal-response of circulating cardiometabolic markers, bile acids and gut hormone as well as calculated insulin sensitivity/secretion. The surgery group patients will undergo surgery as per standard practice and will be reviewed in the bariatric clinic 4-6 weeks' post surgery- this will be at 5-7% weight loss (WL). At the 5-7% WL visit the patient will undergo a metabolic lab panel, a liver FNA, will have their weight and height recorded and BMI calculated. A new FibroScan will be performed.

Additionally, a saliva swab, urine and stool sample will be collected. The 12 patients ( 6 RYGB, 6 SG) in the surgery group who were included in the previous MMT will undergo a second MMT to investigate the change in meal-response of circulating cardio-metabolic markers, bile acids, gut hormones, insulin sensitivity/secretion post-surgery.

The lifestyle intervention group participants will attend a one-to-one dietary consultation with a registered dietician to select a diet plan: either a low-calorie diet or meal replacement diet to induce 5-7% WL. Information booklets that will aid dieting will be provided to the participant. The participant will then be expected to follow the dietary advice in order to achieve a 5-7% WL. The clinical research team will provide additional phone call consultations at 2-, 4-, 8-, 12-, 14-, 16-, 18-, 20-, 22-, 24-weeks post-lifestyle intervention to assess weight change, diet adherence and motivation. Once the participant has a 5-7% WL they will attend the bariatric clinic for their 5-7% WL visit. At the 5-7% WL visit the patient will undergo a metabolic lab panel, a liver FNA, will have their weight and height recorded and BMI calculated. A new FibroScan will be performed. Additionally, a saliva swab, urine and stool sample will be collected. The 6 patients in the lifestyle intervention group who were included in the previous MMT will undergo a second MMT to investigate the change in meal-response of circulating cardio-metabolic markers, bile acids, gut hormones, insulin sensitivity/secretion post-lifestyle intervention.

The outcome measures above will be measured at two time-points; baseline and after 5-7% weight loss in both groups. The study design allows to control for weight loss (through an equivalent weight loss of 5-7% between the two groups) and to understand the effects bariatric/metabolic surgery versus lifestyle intervention (diet and exercise), by mechanisms independent of weight-loss, on markers of NASH and cardiovascular risk, therefore allowing to identify weight-independent effects of bariatric/metabolic surgery, if they exist. Based on published data it is predicted that it will take 3-6 months for patients to achieve 5-7% weight loss (WL) from the lifestyle intervention used in this study and 4-6 weeks after surgery.

Adipose and liver tissue from intraoperative biopsies and gastric and intestinal tissue from surgical waste will be collected and stored for future ethically approved research.

ELIGIBILITY:
Inclusion Criteria:

• BMI greater than 35 kg/m2 (or >32.5. kg/m2 for patients of South Asian, Caribbean or Black ethnicities) with raised alanine transaminase (ALT), aspartate transaminase (AST) and a FibroScan® score > 7.9 (indicating presence of NAFLD and high likelihood of NASH).

Exclusion Criteria:

* other causes of liver disease such as viral, alcoholic (alcohol consumption >20 g/day for women or >30 g/day for men),
* auto-immune disease
* use of certain medications that may interfere with outcome measures (i.e. corticosteroids, insulin and glycoprotein-1 (GLP-1) analogues).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of liver inflammation and fibrosis | Change from baseline to 4-6 weeks (for the surgery group) and to 6 months (lifestyle intervention group)
  Markers of liver injury in blood [i.e. CK-18, tissue inhibitor of metalloproteinases (TIMP-1) amino-terminal pro-peptide of type III collagen (PIIINP), hyaluronic acid].
Assessment of liver inflammation and fibrosis | Change from baseline to 4-6 weeks (for the surgery group) and to 6 months (lifestyle intervention group)
  Serum adipokines [i.e. adiponectin, visfatin, IL-6, TNFa].
Assessment of liver inflammation and fibrosis | Change from baseline to 4-6 weeks (for the surgery group) and to 6 months (lifestyle intervention group)
  FibroScan® score
Assessment of liver inflammation and fibrosis | Change from baseline to 4-6 weeks (for the surgery group) and to 6 months (lifestyle intervention group)
  Fine Needle Aspiration of the liver to obtain a measurement of inflammatory cells in liver

SECONDARY OUTCOMES:
Assessment of markers of cardiovascular disease in fasting and postprandial phase in response to a mixed meal test (MMT) in a subset of patients (total no.=18; 6 RYGB, 6 SG, 6 lifestyle intervention) | Changes from 0 to 30 and 60 minutes after meal consumption.
  Serum levels of apoprotein (apolipoproteins; apoprotein C3, apoprotein C2, and apoprotein E). Blood will be obtained at 0, 30 and 60 minutes.
  • Bile acids: Blood will be obtained at 0, 30 and 60 minutes. Adipose and liver tissue from intraoperative biopsies; gastric and intestinal tissue from surgical waste will be collected. Furthermore, urine, saliva and stool will be obtained at baseline and at 5-7% WL to be stored for use in future downstream hypothesis.
Assessment of gut hormones in fasting and postprandial phase in response to a mixed meal test (MMT) in a subset of patients (total no.=18; 6 RYGB, 6 SG, 6 lifestyle intervention) | Changes from -10 minutes to 0, 15, 30, 60, 90, 120 and 180 minutes after meal consumption.
  Plasma levels gut hormones [i.e.GLP-1, PYY3-36, ghrelin, glucose, insulin, c-peptide levels] will be measured.
Assessment of insulin sensitivity in fasting and postprandial phase in response to a mixed meal test (MMT) in a subset of patients (total no.=18; 6 RYGB, 6 SG, 6 lifestyle intervention) | Changes from -10 minutes to 0, 15, 30, 60, 90, 120 and 180 minutes after meal consumption.
  Oral glucose insulin sensitivity (OGIS) index will be used to calculate insulin sensitivity.
Assessment of bile acids in fasting and postprandial phase in response to a mixed meal test (MMT) in a subset of patients (total no.=18; 6 RYGB, 6 SG, 6 lifestyle intervention) | Changes from 0 to 30 and 60 minutes after meal consumption.
  Measurement of bile acids in blood.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287
- [Background] Rubino F, Nathan DM, Eckel RH, Schauer PR, Alberti KG, Zimmet PZ, Del Prato S, Ji L, Sadikot SM, Herman WH, Amiel SA, Kaplan LM, Taroncher-Oldenburg G, Cummings DE; Delegates of the 2nd Diabetes Surgery Summit. Metabolic Surgery in the Treatment Algorithm for Type 2 Diabetes: A Joint Statement by International Diabetes Organizations. Diabetes Care. 2016 Jun;39(6):861-77. doi: 10.2337/dc16-0236. PMID 27222544
- [Background] Jennings A, Hughes CA, Kumaravel B, Bachmann MO, Steel N, Capehorn M, Cheema K. Evaluation of a multidisciplinary Tier 3 weight management service for adults with morbid obesity, or obesity and comorbidities, based in primary care. Clin Obes. 2014 Oct;4(5):254-66. doi: 10.1111/cob.12066. Epub 2014 Jul 1. PMID 25825858
- [Background] Pembroke T, Gallimore A, Godkin A. Tracking the kinetics of intrahepatic immune responses by repeated fine needle aspiration of the liver. J Immunol Methods. 2015 Sep;424:131-5. doi: 10.1016/j.jim.2015.04.011. Epub 2015 Apr 22. PMID 25914090
- [Background] Pechlaner R, Tsimikas S, Yin X, Willeit P, Baig F, Santer P, Oberhollenzer F, Egger G, Witztum JL, Alexander VJ, Willeit J, Kiechl S, Mayr M. Very-Low-Density Lipoprotein-Associated Apolipoproteins Predict Cardiovascular Events and Are Lowered by Inhibition of APOC-III. J Am Coll Cardiol. 2017 Feb 21;69(7):789-800. doi: 10.1016/j.jacc.2016.11.065. PMID 28209220
- [Background] Halperin F, Ding SA, Simonson DC, Panosian J, Goebel-Fabbri A, Wewalka M, Hamdy O, Abrahamson M, Clancy K, Foster K, Lautz D, Vernon A, Goldfine AB. Roux-en-Y gastric bypass surgery or lifestyle with intensive medical management in patients with type 2 diabetes: feasibility and 1-year results of a randomized clinical trial. JAMA Surg. 2014 Jul;149(7):716-26. doi: 10.1001/jamasurg.2014.514. PMID 24899464
- [Background] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783